CLINICAL TRIAL: NCT01396915
Title: Effects of Increased, Egg-Based Protein Intake on Muscle Composition,
Acronym: S25
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph.D, Purdue University
Other Study IDs: 1101010282
Record Dates: First submitted 2011-02-11; First posted 2011-07-19 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2013-05

CONDITIONS: Muscle Composition; Sarcopenia; Hypertrophy; Inflammation
Keywords: Skeletal muscle lipid content; whole muscle volume; fasting glucose; insulin; blood urea nitrogen
MeSH Terms: conditions — Sarcopenia; Hypertrophy; Inflammation; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood, serum, and muscle tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High or Normal Dietary Protein Intake
  Interventions: Dietary Supplement: Dietary Protein Intake

INTERVENTIONS:
Dietary Supplement: Dietary Protein Intake — Dietary Protein Intake This is a 12-week randomized,prospective study incorporating a dietary intervention in which subjects will consume either higher protein(HP:1.4g protein•kg-1•d-1) or normal protein diet (NP:.8g protein•kg-1•d-1)

SUMMARY:
This study is designed to assess the effect of a diet-controlled nutrition program utilizing an egg-based higher protein diet on muscle composition and size, and indices of metabolic health and markers of systemic inflammation in older men and women who are slightly overweight.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women between the ages of 55-80
* Body Mass Index between 27-35
* Non Diabetic
* Normal liver, kidney and heart functions within 10% of clinical normalcy
* Not currently following a weight loss or other special /non balanced diets
* weight stable

Exclusion Criteria:

* fasting glucose > 110 mg/dl
* blood pressure > 160/110 mm Hg
* plasma total cholesterol > 260 mg/dl
* LDL-cholesterol >160mg/dl
* triacylglycerol>400 mg/dl
* >than 1 hour/week of habitual aerobic and /or resistance exercise
* Currently taking prescribed blood thinners

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and Women between the ages of 65-80
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Effects of Increased, Egg-Based Protein Intake on Muscle Composition, Metabolic Health and Systemic Inflammation in Obese, Older Adults | December 31, 2013
  Anticipated subject recruitment completion

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States